CLINICAL TRIAL: NCT00299117
Title: Effect of a Brief Preoperative Smoking Intervention on Postoperative Complications in Women Undergoing Breast Cancer Surgery: A Randomised Clinical Trial
Brief Title: Brief Smoking Intervention for Women Undergoing Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Ann M. Møller, Research and Development Unit, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KA-20060007
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer; Smoking
Keywords: Smoking cessation; Stress; Nicotine dependence; Complication, postoperative
MeSH Terms: conditions — Breast Neoplasms; Smoking; Smoking Cessation; Tobacco Use Disorder; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Brief preoperative smoking intervention — One counseling session of approximately 45 minutes duration 3-4 days preoperatively. The intervention is inspired by the principles of motivational interviewing and The Stages of Change Model.

SUMMARY:
The primary purpose of this study is to examine the effect of a brief preoperative smoking intervention on postoperative complications in women undergoing breast cancer surgery.

Secondary purposes are to examine long-term smoking cessation rates and experienced stress and nicotine withdrawal symptoms during the smoking cessation period.

DETAILED DESCRIPTION:
Smokers are at greater risk of developing postoperative complications. The connection between smoking and cardiovascular and pulmonary disease is furthermore well documented.

Smoking cessation 6 weeks before orthopaedic surgery significantly reduces the risk of developing postoperative complications. However, smoking cessation for an even shorter period may theoretically have similar effects on postoperative complications.

Intensive smoking intervention programmes increase long-term smoking cessation rates significantly. Little evidence is available on the efficacy of brief smoking intervention programmes for newly diagnosed cancer patients.

This study therefore aims to examine the effect of a brief smoking intervention on postoperative complications and long-term smoking cessation rates in women undergoing breast cancer surgery.

The study is a randomised clinical trial in which study participants are randomised by block randomisation to either standard care (control group) or a brief preoperative smoking intervention (intervention group). Patients in the intervention group are counselled to comply with an intended perioperative smoking cessation period of 13 days.

The intervention and control groups will be compared up to 12 months postoperatively in regard to frequency of postoperative complications and smoking cessation rates. Additionally, experienced stress and nicotine withdrawal symptoms during the perioperative smoking cessation period will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Scheduled for elective breast cancer surgery
* Daily smoker
* Age 18 years and above
* Able to read and write Danish
* Informed consent.

Exclusion Criteria:

* Alcohol intake >35 units per week
* Diagnosed psychiatric disease (including substance abuse and dementia)
* ASA IV and V
* Preoperative neo-adjuvant chemotherapy
* Ulcerating cancer
* Pregnancy and breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Postoperative complications requiring treatment | 6 months postoperatively

SECONDARY OUTCOMES:
Smoking cessation rates | 12 months postoperatively
Experienced stress and nicotine withdrawal symptoms | 10 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, MD, PhD, Study Chair — WHO Collaborating Centre for Evidence-Based Health Promotion Hospitals
Locations (3):
- Denmark (3):
  - Brystkirurgisk Afdeling, Rigshospitalet, Copenhagen, Copenhagen
  - Brystkirurgisk Afdeling, Amtssygehuset i Herlev, Copenhagen, Herlev
  - Ringsted Sygehus, Ringsted, Ringsted